CLINICAL TRIAL: NCT01597596
Title: A Phase 3/4, Prospective, Multinational, Open-label, Noninferiority Study of Alglucosidase Alfa Manufactured at the 160 L and 4000 L Scales in Treatment Naïve Patients With Infantile-Onset Pompe Disease
Brief Title: A Noninferiority Study of Alglucosidase Alfa Manufactured at the 160 L and 4000 L Scales in Treatment Naïve Patients With Infantile-Onset Pompe Disease
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was stopped due to approved label expansion of alglucosidase alfa.
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGLU07510; 2011-005595-42 (EudraCT Number)
Record Dates: First submitted 2012-05-10; First posted 2012-05-14 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-12

CONDITIONS: Pompe Disease (Infantile-Onset); Glycogen Storage Disease Type II (GSD II); Glycogenosis 2; Acid Maltase Deficiency
MeSH Terms: conditions — Glycogen Storage Disease Type II | interventions — GAA protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alglucosidase Alfa 4000 L material (Non-US participants) (Experimental): Alglucosidase alfa 4000 L material for 52 weeks.
  Interventions: Biological: alglucosidase alfa
- Alglucosidase Alfa 160 L material (US participants) (Active Comparator): Alglucosidase alfa 160 L material for 52 weeks.
  Interventions: Biological: alglucosidase alfa

INTERVENTIONS:
Biological: alglucosidase alfa — Intravenous (IV) infusion of alglucosidase alfa (4000 L material) 20 mg/kg every other week (QOW)
  Other Names: Lumizyme
  Arms: Alglucosidase Alfa 4000 L material (Non-US participants)
Biological: alglucosidase alfa — IV infusion of alglucosidase alfa (160 L material) 20 mg/kg QOW.
  Other Names: Myozyme
  Arms: Alglucosidase Alfa 160 L material (US participants)

SUMMARY:
A study to demonstrate comparable safety, efficacy, and pharmacokinetics (PK) of alglucosidase alfa manufactured at the 160 litre (L) and 4000 L scales in participants who had been diagnosed with infantile-onset Pompe disease. Participants were treated with alglucosidase alfa 160 L scale product in the United States (US) and 4000 L scale product in the regions outside the US.

ELIGIBILITY:
Inclusion Criteria:

* The participant's parent/legal guardian was willing and able to provide signed informed consent.
* The participant might be less than or equal to 12 months of age.
* The participant might have documented GAA enzyme deficiency from blood, skin, or muscle tissue.
* The participant might be naïve to treatment with alglucosidase alfa.

Exclusion Criteria:

* The participant was cross-reactive immunologic material negative.
* The participant required invasive ventilator support at the time of enrollment.
* The participant had decompensated clinical heart failure.
* The participant had a major congenital abnormality, excluding cardiac hypertrophy.
* The participant had a clinically significant organ disease (excluding the signs and symptoms of Pompe disease).
* The participant was currently receiving any investigational product.
* The participant was participating in another clinical study.
* The participant and/or the patient's parent/legal guardian was unable to adhere to the requirements of the study.

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (17):
- United States (14):
  - Little Rock, Arkansas
  - Oakland, California
  - Gainsville, Florida
  - Decatur, Georgia
  - Chicago, Illinois
  - Cambridge, Massachusetts
  - Detroit, Michigan
  - Las Vegas, Nevada
  - New Brunswick, New Jersey
  - New York, New York
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Fort Worth, Texas
  - Seattle, Washington
- Germany (2):
  - Geiben
  - Mainz
- Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between 21 August 2012 and 1 December 2014.
Pre-assignment Details: A total of 5 participants were screened and 4 participants were treated.
Groups:
- Alglucosidase Alfa 4000 L Material (Non-US Participants): Alglucosidase alfa (4000 L material) 20 mg/kg intravenous (IV) infusion every other week (QOW) for 52 weeks.
- Alglucosidase Alfa 160 L Material (US Participants): Alglucosidase alfa (160 L material) 20 mg/kg IV infusion QOW for 52 weeks.
Period: Overall Study
Arm/Group | Alglucosidase Alfa 4000 L Material (Non-US Participants) | Alglucosidase Alfa 160 L Material (US Participants)
Started | 1 | 3
Completed | 0 | 2
Not Completed | 1 | 1
Not completed — Study terminated by sponsor | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Alglucosidase Alfa 4000 L Material (Non-US Participants): Alglucosidase alfa (4000 L material) 20 mg/kg IV infusion QOW for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | Alglucosidase Alfa 4000 L Material (Non-US Participants) | Alglucosidase Alfa 160 L Material (US Participants) | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.3 | 0.5 (0.28) | 0.4 (0.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cardiac Function at Week 52
Description: Cardiac function was measured by the left ventricular mass Z-score (LVM-Z). Z-Scores indicate the number of standard deviations (SD) from the mean in a normal distribution. A negative change from baseline indicates a decrease and positive change from baseline indicates an increase in LVM Z-score. The normal range is -2 to 2 and greater than 2 may indicate left ventricular hypertrophy.
Time Frame: Baseline, Week 52
Population: Full analysis population defined as all participants who receive at least 1 infusion of alglucosidase alfa. For this endpoint no participants were analyzed in 'Algucosidase Alfa 4000 L material' arm at Baseline and Week 52. One participant from 'Algucosidase Alfa 160 L Material' arm was discontinued from study at Week 31 due to physician's decision
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Alglucosidase Alfa 4000 L Material (Non-US Participants) | Alglucosidase Alfa 160 L Material (US Participants)
Number analyzed (Participants) | 0 | 2
Z-score |  | -5.06 (1.103)

2. Secondary Outcome: Percentage of Participants With Estimated Probability of Survival
Time Frame: Up to Week 52
Population: Full analysis population.
Measure: Number; unit: percentage of participants
Arm/Group | Alglucosidase Alfa 4000 L Material (Non-US Participants) | Alglucosidase Alfa 160 L Material (US Participants)
Number analyzed (Participants) | 1 | 3
percentage of participants | 100 | 100

3. Secondary Outcome: Number of Participants With Invasive Ventilator-Free Survival
Description: Invasive ventilator-free survival was defined as the time during which the participant is alive and not invasively ventilated. Number of Participants with invasive ventilator-free survival were reported.
Time Frame: Up to Week 52
Population: Full analysis population.
Measure: Number; unit: participants
Arm/Group | Alglucosidase Alfa 4000 L Material (Non-US Participants) | Alglucosidase Alfa 160 L Material (US Participants)
Number analyzed (Participants) | 1 | 3
participants | 1 | 2

4. Secondary Outcome: Change From Baseline in Motor Development Status at Week 52
Description: Motor development status was assessed by the Gross Motor Function Measure - 88 Scale (GMFM-88) total percent scores. GMFM-88 is an 88-item measure to detect gross motor function. It consists of 5 categories: lying and rolling; sitting; crawling and kneeling; standing; walking, running and jumping. Each item was scored on a 4-point Likert scale (0 = cannot do; 1 = initiates [<10% of the task]; 2 = partially completes [10% to <100% of the task]; 3 = task completion). The score for each dimension was expressed as a percentage of the maximum score for that dimension. Total score ranges from 0% to 100%, where higher scores indicate better motor functions.
Time Frame: Baseline, Week 52
Population: Full analysis population. For this endpoint no participants were analyzed in 'Algucosidase Alfa 4000 L material' arm at Baseline and Week 52. One participant from 'Algucosidase Alfa 160 L Material' arm was discontinued from study at Week 31 due to physician's decision.
Measure: Mean (Standard Deviation); unit: percentage of maximum total score
Arm/Group | Alglucosidase Alfa 4000 L Material (Non-US Participants) | Alglucosidase Alfa 160 L Material (US Participants)
Number analyzed (Participants) | 0 | 2
percentage of maximum total score |  | 48.65 (17.183)

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 52) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (the period from the first infusion date to the date that the last data were collected). Analysis was carried out on full analysis population.
Arm/Group | Alglucosidase Alfa 4000 L Material (Non-US Participants) | Alglucosidase Alfa 160 L Material (US Participants)
Serious Adverse Events (participants affected / at risk) | 0/1 | 3/3
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alglucosidase Alfa 4000 L Material (Non-US Participants) (N=1) | Alglucosidase Alfa 160 L Material (US Participants) (N=3)
Cardiac failure (Cardiac disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Adenovirus infection (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Hypotonia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alglucosidase Alfa 4000 L Material (Non-US Participants) (N=1) | Alglucosidase Alfa 160 L Material (US Participants) (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Nodal rhythm (Cardiac disorders) | 0 | 1
Middle ear effusion (Ear and labyrinth disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Device occlusion (General disorders) | 0 | 1
Infusion site erythema (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 3
Bronchitis (Infections and infestations) | 0 | 1
Croup infectious (Infections and infestations) | 0 | 1
Eye infection (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.